CLINICAL TRIAL: NCT07296484
Title: Clofutriben And Placebo Phase 2 Trial Against INtractable Type 2 Diabetes (CAPTAIN-T2D)
Brief Title: Trial Against INtractable Type 2 Diabetes (CAPTAIN-T2D)
Acronym: CAPTAIN-T2D
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SPI-62-CL-2006
Record Dates: First submitted 2025-11-30; First posted 2025-12-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes; Cortisol Excess
Keywords: hypercortisolism; Cortisol excess; elevated cortisol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; ACTH Syndrome, Ectopic; Cushing Syndrome | interventions — ASP3662

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose 1 (Experimental): clofutriben .2 mg oral tablet daily
  Interventions: Drug: clofutriben
- Dose 2 (Experimental): clofutriben 2mg oral tablet daily
  Interventions: Drug: clofutriben
- Dose 3 (Experimental): clofutriben 6mg oral tablet daily
  Interventions: Drug: clofutriben
- Dose 4 (Experimental): clofutriben 12 mg oral tablet daily
  Interventions: Drug: clofutriben
- placebo (Placebo Comparator): placebo control oral tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: clofutriben — HSD-1 inhibitor
  Other Names: SPI-62; ASP3662
  Arms: Dose 1; Dose 2; Dose 3; Dose 4
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
CAPTAIN-T2D will take place in two parts. Part 1 (Screening) will evaluate patients with type 2 diabetes and elevated cortisol risk factors for trial eligibility and the presence of elevated cortisol. Participants deemed eligible from Part 1 will be randomized to either clofutriben or placebo in the double-blind (participant and investigator), dose-ranging, interventional Part 2 (Treatment).

DETAILED DESCRIPTION:
CAPTAIN-T2D is a two-part, multicenter, randomized, double-blind, parallel group, placebo- controlled trial of the 11-hydroxysteroid dehydrogenase type 1 (HSD-1) inhibitor clofutriben. The primary objectives of this trial are to characterize the relationship of clofutriben dose to improved glycemic control, and to identify one or more doses suitable for Phase 3 evaluation, in patients with T2D and elevated cortisol.

The trial consists of two parts.

Part 1 (Screening) will last between approximately 5 to 9 weeks for most participants. The screening period duration allows for (sequentially) initial eligibility screen, dexamethasone suppression test, and further eligibility assessments.

During Part 2 (Treatment), participants will be randomized to placebo or one of four clofutriben doses. Part 2 will last 24 weeks with a follow-up phone call 4 weeks after the last dose of trial medication.

ELIGIBILITY:
Inclusion Criteria:

* From Screening 1

  * Age at least 18 years.
  * HbA1c ≥7.5% documented within 3 months prior to Screening 1. (The historical HbA1c value must have been obtained after at least 2 months on the current [as of Screening 1] regimen).
  * Treatment with stable and adequate doses of ≥2 injectable or oral ADMs. (An ADM will be deemed stable if the dose has been the same for at least 3 months prior to Screening 1 and without change between Screening 1 and Day 1) (An ADM dose will be deemed adequate if it is at or above the maximal labelled dose, or a sub-maximal, but not starting, dose if limited by tolerability (confer with MM if less than half-maximal dose).
  * Adequate total daily insulin is defined as at least 0.3 units/kg/day. Insulin dose will be deemed stable with adjustments of up to 20% total daily dose during the 3 months prior to Screening 1 or between Screening 1 and Day 1.
  * Use of insulin pumps or insulin brand changes (e.g., due to insurance change or shortage) are to be discussed with the MM.
  * At least one of the following

    * ≥3 stable and adequate ADMs;
    * diabetes complication (retinopathy, nephropathy, neuropathy, atherosclerotic heart disease);
    * hypertension requiring ≥2 adequately dosed AHMs;
    * adequately dosed basal or basal plus prandial insulin in addition to at least 1 other ADM; and
    * adequately dosed incretin agonist (a single or combination agent counts as one ADM) in addition to at least 1 other ADM;
    * evidence or history of osteoporosis or non-traumatic fracture (e.g., vertebral body compression);
    * or established diagnosis of a neoplastic (non-malignant) source of hypercortisolism and have failed, are ineligible for, or declined surgery.

At DST • Post-DST cortisol level >1.8 µg/dL and serum dexamethasone ≥140 ng/dL. Patients with an established diagnosis of neoplastic hypercortisolism do not require a DST.

At Screening 2

* HbA1c ≥7.5% at Screening 2. At Day 1
* No change in, or initiation of, medications for hypertension within 1 month prior to Day 1.

Exclusion Criteria:

* New-onset diabetes (onset <1 year in the past).
* Unwillingness to maintain with current glucose-lowering regimen during the trial.
* Unwillingness to adjust, add, replace, or discontinue current or other glucose-lowering medications during the trial as directed by the investigator.
* Unwillingness to comply with CGM or other trial procedures.
* Investigator considers the patient will otherwise be unwilling or unable to complete the trial.
* Night-shift worker or otherwise habitually awake from 23:00 to 07:00 h.
* Evidence for significant hypoglycemia while on their current diabetic treatment regimen(This includes episodes of symptomatic Level 3 hypoglycemia requiring external assistance for recovery, or CGM-documented prolonged [>15 min] or repeated episodes of either Level 2 hypoglycemia leading to >1%, or Level 1 hypoglycemia leading to >4%, in "time below range" within 3 months prior to Screening 1 or between Screening 1 and Day 1).
* Any of the following in medical history:

  * Type 1 diabetes mellitus (T1D), latent autoimmune diabetes in adults (LADA), or familial forms of maturity-onset diabetes of the young (MODY);
  * A hemoglobinopathy or other condition which may interfere with measurement of HbA1c (e.g., sickle cell disease HbSS or other variants HbEE thalassemia, hemolytic anemia, recent blood transfusion);
  * Hypersensitivity or severe reaction to dexamethasone;
  * Pheochromocytoma, or suspicion thereof;
  * Anorexia, or other eating disorder;
  * Glucocorticoid resistance;
  * Multiple sclerosis;
  * Significant hepatic impairment (e.g., Child-Pugh Class B or C);
  * Idiopathic thrombocytopenic purpura;
  * Untreated or inadequately controlled moderate-to-severe sleep apnea (apnea-hypopnea index ≥15). (Patients whose condition has been well controlled with Continuous Positive Airway Pressure (CPAP) use for at least 3 months prior to Screening 1 are not excluded. Patients with a STOP-BANG score 5-8 should be referred for a sleep study outside the trial and may rescreen if found not to have moderate-to-severe sleep apnea);
  * Current alcohol consumption >14 units/week or >4 units in a single day for males, or >7 units/week or >3 units in a single day for females. (Patients with a CAGE score 2-4 should be evaluated further outside the trial and may be rescreened if found not to have an alcohol [or other substance] use disorder);
  * Untreated or inadequately controlled major depressive disorder, generalized anxiety disorder, bipolar disorder, post-traumatic stress disorder, or schizophrenia.(Patients whose condition has been well controlled with stable medical therapy, or has been asymptomatic, for at least 3 months prior to Screening 1 are not excluded); or
  * Any other medical condition (including malignancy) that is likely to interfere with trial assessments or the patient's ability to complete the trial.
  * Any of the following in medication history:
  * Any of the excluded medications listed in Section 6.9;
  * Any investigational drug within 4 weeks or within less than five times the drug's half-life, whichever is longer, prior to Screening 1 or between Screening 1 and Day 1;
  * Woman of childbearing potential (WOCBP) not willing to adhere to highly effective contraception or strict abstinence for the duration of the trial and for 90 days post completion/discontinuation; and
  * Pregnancy (including a positive urine test) or current breast feeding.

From Screening 2

• Prior probability of undiagnosed endogenous Cushing syndrome based on either of:

* wo morning serum cortisol values after dexamethasone suppression >5.0 mcg/dL together with plasma dexamethasone >140 ng/mL; or
* a morning serum cortisol value after dexamethasone suppression >1.8 mcg/dL, together with plasma dexamethasone >140 ng/mL and any one of the following that is not attributable to an etiology other than endogenous Cushing's syndrome:
* supraclavicular/dorsocervical fat accumulation;
* irounding of the face (especially compared with prior photos);
* skin changes (violaceous striae, skin thinning, or excessive bruising);
* proximal muscle weakness on exam; or
* history of deep vein thrombosis/pulmonary embolism.
* Plans for, or medically unable to forego, treatment for endogenous Cushing syndrome or ACS within the next 8 months. (For clarity, patients with EnCS or ACS, not having such treatment plans, and medically able to forego treatment for 8 months may enroll if otherwise eligible).
* Severe, poorly controlled hypertension (mean systolic BP >160 mmHg or mean diastolic BP >100 mmHg) at Screening 2 or between Screening 2 and Day 1, including by at-home monitoring. (Such patients will be eligible to rescreen for Part 2 when they restore BP <160/100 mmHg for 1 month on a new stable medication regimen).
* Positive urine screen for recreational drugs (except tetrahydrocannabinol (THC)).
* Glomerular filtration rate (GFR) (determined using Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) <45 mL/min/1.73 m².
* Poorly controlled hyperthyroidism/hypothyroidism (confirmed by TSH or Free thyroxine [fT4]).
* Liver enzymes >3 × upper limit of normal (ULN) (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or bilirubin >1.5 × ULN.(excepting benign conditions such as Gilbert's)
* Known hypersensitivity to clofutriben or to any of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with both morning serum cortisol >1.8 mg/dL and morning plasma dexamethasone >=140 ng/dL (single composite endpoint) after a single dexamethasone 1 mg dose taken the prior night. | 8-10 hours after the dexamethasone 1 mg dose.
  To assess prevalence in the trial population of morning cortisol non-suppression by a single dexamethasone 1 mg dose.
Glycated hemoglobin A1c (%) change from baseline to Week 24 by treatment. | 24 weeks.
  To assess glycated hemoglobin A1c (%) changes, compared to placebo, in patients who receive each of 4 daily clofutriben doses for 24 weeks.

SECONDARY OUTCOMES:
Fasting plasma glucose (mmol/L) change from baseline to Week 24 by treatment. | 24 weeks
  To assess glucose (mmol/L) changes, compared to placebo, in patients who receive each of 4 daily clofutriben doses for 24 weeks.

OTHER OUTCOMES:
To evaluate the safety of clofutriben in participants with T2D and EC. | From enrollment until end of trial 9 month
  Frequency of TEAEs (treatment-emergent adverse even) by clofutriben dose

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Arizona Clinical Trials - Pecos, Chandler, Arizona
  - Arizona Clinical Trials - Broadway, Tucson, Arizona
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research - Gardena, La Mesa, California
  - Ark Clinical Research - Long Beach, Long Beach, California
  - Los Angeles Institute for Metabolic Research, Los Angeles, California
  - Velocity Clinical Research, Los Angeles, Los Angeles, California
  - Amicis Research Center- Nordhoff, Northridge, California
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Admed Research LLC, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - IACT Health-Brookstone Centre Pkwy, Columbus, Georgia
  - Chicago Clinical Research Institute, Chicago, Illinois
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - NOLA Care Clinical Research, Metairie, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Medstar Health Research Institute, Olney, Maryland
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Oakland Medical Research Center, Troy, Michigan
  - Velocity Clinical Research, Lincoln, Lincoln, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Velocity Clinical Research, Binghamton, Binghamton, New York
  - Endocrine Associates of Long Island, P.C., Smithtown, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Physicians East, Greenville, North Carolina
  - Lucas Research Inc, Morehead City, North Carolina
  - Velocity Clinical Research, Cincinnati, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Blue Ash, Cincinnati, Ohio
  - Endocrinology Associates, Inc, Columbus, Ohio
  - Remington Davis, Inc, Columbus, Ohio
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - Velocity Clinical Research, Austin, Austin, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - Juno Research, LLC, Houston, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - Texas Diabetes & Endocrinology, P.A. - Round Rock, Round Rock, Texas
  - Elevate Clinical Research, Seabrook, Texas
  - Texas Valley Clinical Research, LLC, Weslaco, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Velocity Clinical Research, Suffolk, Suffolk, Virginia